CLINICAL TRIAL: NCT00671775
Title: Cognitive Effects of Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Columbia University (Other); Weill Medical College of Cornell University (Other); Kent State University (Other); Neuropsychiatric Research Institute, Fargo, North Dakota (Other)
Responsible Party: Sponsor
Other Study IDs: DK75119; R01DK075119 (NIH)
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Bariatric Surgery Patients
Keywords: Bariatric Surgery; Obesity; Cognitive Function
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Bariatric surgery patients
- Weight loss programs

SUMMARY:
There is growing evidence that obesity is associated with adverse neurocognitive outcome. Recent studies demonstrate that elevated body mass index (BMI) is an independent risk factor for Alzheimer's disease, structural brain abnormalities, and cognitive dysfunction in older adults. Preliminary work from our lab extends these findings and shows structural brain differences and cognitive dysfunction also exist in obese young and middle-aged adults.

Bariatric surgery is increasingly viewed as an effective intervention for morbid obesity, though its effects on cognition are unknown. Post-operative nutritional deficiencies are common and can adversely impact cognitive performance. However, substantial weight loss resolves or improves many medical conditions with reversible cognitive effects, suggesting bariatric surgery may provide cognitive benefits.

No study to date has examined the cognitive effects of bariatric surgery. To do so, the proposed study will prospectively assess cognitive performance in 125 bariatric surgery patients enrolled in the Longitudinal Assessment of Bariatric Surgery (LABS) project and 125 matched controls. Bariatric surgery patients will complete a computerized cognitive test battery at four time points: pre-operatively, 12 weeks post-operatively, 12 months post-operatively, and 24 months post-operatively. Matched control participants will complete the test battery at similar intervals. Demographic, medical, and psychosocial information will be collected to elucidate possible mechanisms of change. We hypothesize that the substantial weight loss following bariatric surgery will be associated with improved cognitive performance.

ELIGIBILITY:
Specific criteria for bariatric surgery patients include:

Inclusion Criteria

* 25-65 years of age
* Enrolled in LABS project
* English-speaking

Exclusion Criteria

* History of neurological disorder or injury (e.g. dementia, stroke, seizures)
* Moderate or severe head injury (defined as >10 minutes loss of consciousness; Alexander, 1995)
* Past or current history of severe psychiatric illness (e.g. schizophrenia, bipolar disorder)
* Past or current history of alcohol or drug abuse (defined by DSM-IV criteria)
* History of learning disorder or developmental disability (defined by DSM-IV criteria)
* Impaired sensory function

Inclusion/exclusion criteria for matched control participants include:

* All of the inclusion/exclusion criteria for the surgical patients, except for enrollment in the LABS project
* No history of bariatric surgery procedures
* No interest in bariatric surgery procedures in the next two years

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the bariatric and weight loss programs of affiliated clinical centers.
Sampling Method: Non-Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Gunstad, Ph.D., Principal Investigator — Kent State University
Locations (1):
- Columbia, New York, New York, United States

REFERENCES:
- [Derived] Garcia S, Fedor A, Spitznagel MB, Strain G, Devlin MJ, Cohen RA, Paul RH, Crosby RD, Mitchell JE, Gunstad J. Patient reports of cognitive problems are not associated with neuropsychological test performance in bariatric surgery candidates. Surg Obes Relat Dis. 2013 Sep-Oct;9(5):797-801. doi: 10.1016/j.soard.2012.10.008. Epub 2012 Oct 30. PMID 23245496